CLINICAL TRIAL: NCT01910311
Title: The Effect of CYP3A Induction by Rifampicin on the Pharmacokinetics of Baricitinib in Healthy Subjects
Brief Title: A Study of Baricitinib and Rifampicin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14608; I4V-MC-JAGK (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): Single oral dose of 10 milligrams (mg) baricitinib on Day 1.
  Interventions: Drug: Baricitinib
- Baricitinib + Rifampicin (Experimental): Oral doses of 600 mg rifampicin once daily on Days 3 to 11, with a single oral dose of 10 mg baricitinib co-administered on Day 10.
  Interventions: Drug: Baricitinib; Drug: Rifampicin

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Rifampicin — Administered orally
  Arms: Baricitinib + Rifampicin

SUMMARY:
The purposes of this study are to look at what effect multiple doses of rifampicin have on a single dose of baricitinib and to look at the safety and tolerability of these drugs. Side effects will be documented. The study will last approximately 31 days from the first dose to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Male participants: Agree to use 2 reliable methods of birth control with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug
* Female participants: Women not of childbearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, bilateral oophorectomy with or without hysterectomy, or bilateral tubal occlusion/ligation) confirmed by medical history, or menopause. Menopausal women are women with spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example, oral contraceptives, hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy). Menopausal status should be confirmed by a follicle-stimulating hormone (FSH) level greater than 40 international units per liter (IU/L) at screening [unless the participant is taking hormone replacement therapy (HRT)]
* Have a body weight of ≥60 kilograms (kg) at the time of screening
* Have clinical laboratory test results within normal reference range
* Have normal renal function
* Have normal blood pressure and pulse rate (supine position)
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Are currently enrolled in, have completed, or discontinued within the last 90 days from a clinical trial involving a study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received the study drug
* Have known allergies to baricitinib, rifampicin, related compounds, or any components of the baricitinib or rifampicin formulations, or history of significant atopy
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption 48 hours prior to the first dose and until completion of the safety follow-up assessment [Day 18 ± 1; 1 unit = 12 ounces (oz) or 360 milliliters (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Have a history of, in the opinion of the investigator, excessive methylxanthine use within previous 6 months, such as greater than (>)6 cups of coffee (or equivalent) per day
* Currently smoke more than 10 cigarettes per day or are unable to abide by Clinical Research Unit (CRU) restrictions
* Are unwilling to refrain from using soft contact lenses from the start of the second treatment period until after the final follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, fixed-sequence, 2-period study conducted in healthy participants to compare the single dose pharmacokinetics (PK) of baricitinib when given alone and when coadministered with rifampicin.
Groups:
- Baricitinib Then Baricitinib and Rifampicin: Period 1: 10-milligram (mg) dose of baricitinib (2 x 4-mg and 1 x 2-mg tablets) administered orally on Day 1.
  Period 2: 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally once daily (QD) on Days 3 through 11, with coadministration of a 10-mg dose of baricitinib on Day 10.
Period: Period 1 (Days 1-2)
Arm/Group | Baricitinib Then Baricitinib and Rifampicin
Started | 18
Received Baricitinib | 18
Completed | 18
Not Completed | 0
Period: Period 2 (Days 3-32)
Arm/Group | Baricitinib Then Baricitinib and Rifampicin
Started | 18
Received Baricitinib | 18
Received At Least 1 Dose of Rifampicin | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib Then Baricitinib and Rifampicin: Period 1: 10-mg dose of baricitinib (2 x 4-mg and 1 x 2-mg tablets) administered orally on Day 1.
  Period 2: 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally QD on Days 3 through 11, with coadministration of a 10-mg dose of baricitinib on Day 10.
Arm/Group | Baricitinib Then Baricitinib and Rifampicin
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: PK: Maximum Concentration (Cmax) of Baricitinib
Time Frame: Period 1, Day 1 and Period 2, Day 10: Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: Participants who received study drug (baricitinib in Period 1 and at least 1 dose of rifampicin and baricitinib in Period 2) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Baricitinib: Period 1: 10-mg dose of baricitinib (2 x 4-mg and 1 x 2-mg tablets) administered orally on Day 1.
- Baricitinib and Rifampicin: Period 2: 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally QD on Days 3 through 11, with coadministration of a 10-mg dose of baricitinib on Day 10.
Arm/Group | Baricitinib | Baricitinib and Rifampicin
Number analyzed (Participants) | 18 | 18
nanograms per milliliter (ng/mL) | 96.1 (22) | 101 (28)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From 0 to Infinity [AUC(0-∞)] of Baricitinib
Time Frame: Period 1, Day 1 and Period 2, Day 10: Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- Baricitinib and Rifampicin: Period 2: 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally QD on Days 3 through 11, with a coadministration of 10-mg dose of baricitinib on Day 10.
Arm/Group | Baricitinib | Baricitinib and Rifampicin
Number analyzed (Participants) | 18 | 18
nanograms*hour/milliliter (ng*h/mL) | 634 (19) | 416 (20)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Baricitinib
Time Frame: Period 1, Day 1 and Period 2, Day 10: Predose, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: Participants who received study drug (baricitinib in Period 1 and at least 1 dose of rifampicin and baricitinib in Period 2) and who had evaluable PK data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Baricitinib | Baricitinib and Rifampicin
Number analyzed (Participants) | 18 | 18
hours (h) | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.00]

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 32)
Groups:
- Baricitinib: A 10-mg dose of baricitinib (2 x 4-mg and 1 x 2-mg tablets) administered orally on Day 1.
  Adverse events (AEs) are reported from baseline through predose on Day 3.
- Rifampicin: A 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally QD on Days 3 through 9.
  AEs are reported postdose on Day 3 through predose on Day 10.
- Baricitinib and Rifampicin: A 600-mg dose of rifampicin (2 x 300-mg capsules) administered orally QD on Days 10 and 11, with coadministration of a 10-mg dose of baricitinib on Day 10.
  AEs are reported postdose on Day 10 up to Day 32.
Arm/Group | Baricitinib | Rifampicin | Baricitinib and Rifampicin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 3/18 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (N=18) | Rifampicin (N=18) | Baricitinib and Rifampicin (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days